CLINICAL TRIAL: NCT03520920
Title: A Phase 2 Study to Assess the Safety, Tolerability, and Activity of BGB-3111 in Combination With Rituximab in Chinese Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (Non-GCB Subtype) and Relapsed/Refractory Indolent Lymphoma (Follicular Lymphoma and Marginal Zone Lymphoma)
Brief Title: BTK Inhibitor BGB-3111 in Chinese Participants With Diffuse Large B-Cell Lymphoma (Non-GCB) and Indolent Lymphoma (FL and MZL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-213; CTR20170965 (Registry Identifier: China Drug Trials (CDT))
Record Dates: First submitted 2018-04-28; First posted 2018-05-11 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Marginal Zone Lymphoma; Follicular Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R/R Non-GCB DLBCL (Experimental): Participants with non-GCB DLBCL received zanubrutinib plus rituximab for up to progressive disease or intolerance.
  Interventions: Drug: Zanubrutinib; Drug: Rituximab
- R/R FL or MZL (Experimental): Participants with R/R FL or MZL received zanubrutinib plus rituximab for up to progressive disease or intolerance.
  Interventions: Drug: Zanubrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — Administered zanubrutinib 160 mg orally (PO) BID continuously
  Other Names: BGB-3111
Drug: Rituximab — Administered rituximab 375 mg/m^2 intravenously on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.

SUMMARY:
This was a multicenter, open-label, phase 2 study to evaluate efficacy, safety, and tolerability of BGB-3111 (zanubrutinib) 160 milligrams (mg) twice daily (BID) in combination with rituximab in Chinese participants with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) (non-GCB [non-germinal center B-cell-like] subtype) and R/R indolent lymphoma (follicular lymphoma [FL] and marginal zone lymphoma [MZL]).

ELIGIBILITY:
Key Inclusion Criteria:

1. ≥ Age 18 years at time of signing of informed consent.
2. Measurable disease by computed tomography (CT) or positron emission tomography/CT or magnetic resonance imaging, defined as ≥1 nodal lesion that was >1.5 centimeters (cm) in the longest diameter, or ≥1 extra-nodal lesion (for example, hepatic nodules) that was >1 cm in the longest diameter.
3. Availability of archival or fresh tumor tissue sample from an evaluable core or excisional biopsy.
4. Participants meet the following criteria:

   1. Cohort 1: R/R non-GCB DLBCL i. Histologically confirmed non-GCB DLBCL per Hans criteria with non-transformed disease; additional methodologies for confirming non-GCB DLBCL may have been considered in consultation with the medical monitor. ii. Relapsed disease (disease progression after most recent therapy for DLBCL occurring more than 6 months after the completion of last therapy) or refractory disease (failure to achieve complete response [CR] or partial response [PR] to therapy for non-GCB DLBCL or disease progression within 6 months after completion of the most recent therapy for non-GCB DLBCL). iii. Must have received at least one standard anthracycline ± rituximab-based treatment (for example, rituximab plus cyclophosphamide, doxorubicin [or epirubicin, hydroxydaunorubicin, or similar], vincristine, and prednisone) or cyclophosphamide, vincristine, and prednisone +/- rituximab for DLBCL.
   2. Cohort 2: R/R FL or R/R MZL i. Histologically confirmed CD20+ FL (Grade 1, 2, or 3a) or MZL. ii. Relapsed disease (disease progression after most recent therapy for FL or MZL occurring more than 6 months after the completion of last therapy) or refractory disease (failure to achieve complete response (CR) or partial response (PR) to most recent therapy for FL or MZL, or disease progression within 6 months after completion of the most recent therapy for FL or MZL).
5. Laboratory parameters as specified below:

   1. Hematologic: Platelet count ≥75 x 10^9/liter (L) independent of growth factor or transfusion within 7 days of study entry; absolute neutrophil count (ANC) ≥1 x 10^9/L independent of growth factor within 7 days of study entry, hemoglobin >8 grams/deciliter within 7 days of study entry.
   2. Hepatic: Total bilirubin ≤ 2x upper limit of normal (ULN) unless documented Gilbert's syndrome; aspartate aminotransferase/serum glutamic-oxaloacetic transaminase and alanine transaminase/serum glutamic-pyruvic transaminase ≤3x ULN.
   3. Renal: Creatinine clearance ≥30 milliliters/minute (as estimated by the Cockcroft-Gault equation based on ideal body weight or as measured by nuclear medicine scan or 24-hour urine collection).
   4. International normalized ratio and activated partial thromboplastin time ≤1.5x ULN. Participants with anti-phospholipid syndrome, acquired von Willebrand disease, factor inhibitors or on vitamin K antagonist may have been enrolled after discussion with the Medical Monitor.
6. Left ventricular ejection fraction ≥50%.
7. Life expectancy ≥6 months.
8. Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
9. Female participants of childbearing potential must have practiced highly effective methods of contraception initiated prior to first dose of study drug, for the duration of the study, and for ≥90 days after the last dose of zanubrutinib, or 12 months after the last dose of rituximab, whichever is longer.
10. Male participants were eligible if vasectomized or if they agreed to the use of barrier contraception in combination with other methods above during the study treatment period and for ≥90 days after the last dose of zanubrutinib.
11. Able to provide written informed consent and could understand and comply with the requirements of the study.

Key Exclusion Criteria:

1. Known central nervous system lymphoma or leukemia.
2. Histological confirmed gastric mucosa-associated lymphoid tissue type MZL.
3. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
4. Clinically significant cardiovascular disease.
5. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
6. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
7. Severe or debilitating pulmonary disease.
8. Hypersensitivity reaction to zanubrutinib or rituximab or any of the other ingredients of the study drugs.
9. Prior Bruton tyrosine kinase inhibitor treatment.
10. Required ongoing treatment with a strong cytochrome P450 protein inhibitor or inducer.
11. Vaccination with a live vaccine within 28 days of the first dose of study drug.
12. Hematopoietic stem cell transplantation within 6 months of first dose of study drug.
13. Receipt of the following treatment prior to first dose of study drug:

    1. Corticosteroids at doses >20 mg/day prednisone equivalent or steroids given with anti-neoplastic intent within 7 days prior to first dose of study drug.
    2. Chemotherapy or radiotherapy within 4 weeks.
    3. Monoclonal antibody within 4 weeks.
    4. Investigational therapy within 4 weeks.
    5. Chinese patent medicine with anti-neoplastic intent within 4 weeks.
14. Not recovered from toxicity of any prior anti-cancer therapy to ≤Grade 1, except for alopecia, ANC, hemoglobin (Hgb), and platelets. For ANC, Hgb and platelets, see inclusion criterion #5.
15. Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.
16. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, history of bariatric surgery, or partial or complete bowel obstruction.
17. Major surgery within 4 weeks prior to first dose of study treatment.
18. Active fungal, bacterial and/or viral infection requiring systemic therapy.
19. Known infection with human immunodeficiency virus, or serologic status reflecting active hepatitis B or C infection as follows:

    1. Presence of hepatitis B surface antigen (HBsAg) or anti-hepatitis B core antibody (anti-HBc). Participants with presence of anti-HBc, but absence of HBsAg, were eligible if hepatitis B virus (HBV) DNA was <500 international units (IU)/mL, anti-viral therapy started before the first dose of study treatment, and if they were willing to undergo monthly monitoring for HBV reactivation.
    2. Presence of hepatitis C virus (HCV) antibody. Participants with presence of HCV antibody were eligible if HCV RNA was undetectable (<15 IU/mL).
20. Pregnant or lactating women.
21. Underlying medical conditions that, in the investigator's opinion, would have rendered the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
22. Concurrent participation in another therapeutic clinical trial.

Note: Other protocol defined Inclusion/Exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Qingyuan Zhang, Rong Tao, Zhenyu Li, et al. Zanubrutinib (BGB-3111) in combination with rituximab in patients with relapsed/refractory Non-Hodgkin Lymphoma [EHA-2188].

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 study centers in China, all of which enrolled participants. The first enrolled participants received their first dose on 04 January 2018, and the last participant enrolled received their first dose on 20 December 2018. A total of 41 participants with non-Hodgkin lymphoma (NHL) were enrolled into the study, and all received ≥1 dose of study treatment.
Groups:
- Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma: Participants with relapsed/refractory (R/R) non-germinal center B-cell-like diffuse large B-cell lymphoma (non-GCB DLBCL) received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 milligrams (mg) orally (PO) twice daily (BID) continuously and rituximab 375 mg/meter squared (m^2) intravenously (IV) on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Follicular Lymphoma: Participants with R/R follicular lymphoma (FL) received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 IV on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Marginal Zone Lymphoma: Participants with R/R marginal zone lymphoma (MZL) received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 IV on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
Period: Overall Study
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Started | 20 | 16 | 5
Received at Least 1 Dose of Study Drug | 20 | 16 | 5
Completed | 0 | 0 | 0
Not Completed | 20 | 16 | 5
Not completed — Death | 13 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Study Terminated by the Sponsor | 5 | 14 | 5

BASELINE CHARACTERISTICS:
Groups:
- Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma: Participants with R/R non-GCB DLBCL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 IV on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Follicular Lymphoma: Participants with R/R FL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 IV on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Marginal Zone Lymphoma: Participants with R/R MZL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 IV on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Total: Total of all reporting groups
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma | Total
Number analyzed (Participants) | 20 | 16 | 5 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (15.00) | 47.6 (12.36) | 61.2 (8.87) | 53.0 (13.94)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 14 | 15 | 3 | 32
  ≥65 years | 6 | 1 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 3 | 18
  Male | 13 | 8 | 2 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 16 | 5 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kilogram/m^2] | 23.43 (2.652) | 25.04 (5.079) | 24.33 (4.813) | 24.17 (3.989)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.72 (0.113) | 1.77 (0.295) | 1.69 (0.240) | 1.74 (0.213)
Eastern Cooperative Oncology Group Performance (ECOG)Status [Count of Participants; unit: Participants] — ECOG Performance Status - Grade 0 = Fully active, able to carry on all pre-disease performance without restriction; Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; Grade 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    Grade 0 | 13 | 11 | 3 | 27
    Grade 1 | 5 | 4 | 2 | 11
    Grade 2 | 2 | 1 | 0 | 3
Hepatitis B Core Antibody [Count of Participants; unit: Participants]
  Positive | 6 | 3 | 2 | 11
  Negative | 14 | 13 | 2 | 29
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) As Measured By The Investigator
Description: The percentage of participants whose best overall response met partial response (PR) or complete response (CR) criteria among all participants. The 95% confidence interval (CI) was calculated with the Clopper-Pearson method.
Time Frame: Up to approximately 2.5 years
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug (zanubrutinib or rituximab) on the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma: Participants with R/R non-GCB DLBCL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 intravenously on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Follicular Lymphoma: Participants with R/R FL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 intravenously on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
- Relapsed/Refractory Marginal Zone Lymphoma: Participants with R/R MZL received zanubrutinib plus rituximab for up to progressive disease or intolerance. Administered zanubrutinib 160 mg PO BID continuously and rituximab 375 mg/m^2 intravenously on Cycle 1 Days 1, 8, 15, 22, and on Day 1 of Cycles 4, 6, 8, 10. Each cycle was 28 days long.
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Percentage of Participants | 35 [15.4 to 59.2] | 56.3 [29.9 to 80.2] | 60.0 [14.7 to 94.7]

2. Secondary Outcome: Duration Of Response (DOR) As Determined By Investigator
Description: The DOR was defined as the time from the date that the response criteria were first met to the date that progressive disease (PD) was objectively documented or death, whichever occurred first. Medians were estimated by the Kaplan-Meier method with 95% CIs estimated using the Brookmeyer and Crowley method.
Time Frame: Up to approximately 2.5 years
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug (zanubrutinib or rituximab) on the study. Duration of response was summarized for responders (participants with a best response of partial response or higher) only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 7 | 9 | 3
Months | 8.79 [0.72 to NA] — NA = Not estimable due to insufficient number of participants with events | NA [5.45 to NA] — NA = Not estimable due to insufficient number of participants with events | 22.18 [8.31 to NA] — NA = Not estimable due to insufficient number of participants with events

3. Secondary Outcome: DOR: Event-free Rate
Description: The DOR was defined as the time from the date that the response criteria were first met to the date that progressive disease (PD) was objectively documented or death, whichever occurred first. The event-free rate was estimated by the Kaplan-Meier method with 95% CIs estimated using Greenwood's formula.
Time Frame: Up to approximately 2.5 years
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug (zanubrutinib or rituximab).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Percentage of Participants
  6 months | 50.0 [11.1 to 80.4] | 88.9 [43.3 to 98.4] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  9 months | 50.0 [11.1 to 80.4] | 77.8 [36.5 to 93.9] | 66.7 [5.4 to 94.5]
  12 months | 50.0 [11.1 to 80.4] | 64.8 [25.3 to 87.2] | 66.7 [5.4 to 94.5]
  15 months | 33.3 [4.6 to 67.6] | 51.9 [16.4 to 78.8] | 66.7 [5.4 to 94.5]
  18 months | 33.3 [4.6 to 67.6] | 51.9 [16.4 to 78.8] | 66.7 [5.4 to 94.5]
  24 months | NA [NA to NA] — NA = Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA = Not estimable due to insufficient number of participants with events | 33.3 [0.9 to 77.4]

4. Secondary Outcome: Progression-free Survival (PFS) As Determined By Investigator
Description: The PFS was defined as time from first dose of study treatment until first documentation of progression, assessed per the Lugano Classification, or death, whichever occurred first. Medians were estimated by the Kaplan-Meier method with 95% CIs estimated using the Brookmeyer and Crowley method.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Months | 3.38 [2.69 to 5.49] | 11.10 [5.49 to NA] — NA = Not estimable due to insufficient number of participants with events | 24.87 [11.01 to NA] — NA = Not estimable due to insufficient number of participants with events

5. Secondary Outcome: PFS: Event-free Rate
Description: The PFS was defined as time from first dose of study treatment until first documentation of progression, assessed per the Lugano Classification, or death, whichever occurred first. The event-free rate was estimated by the Kaplan-Meier method with 95% CIs estimated using Greenwood's formula.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Percentage of Participants
  6 months | 17.4 [4.3 to 37.7] | 73.3 [43.3 to 89.1] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  9 months | 17.4 [4.3 to 37.7] | 66.7 [37.5 to 84.6] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  12 months | 17.4 [4.3 to 37.7] | 46.7 [21.2 to 68.7] | 80.0 [20.4 to 96.9]
  15 months | 17.4 [4.3 to 37.7] | 46.7 [21.2 to 68.7] | 60.0 [12.6 to 88.2]
  18 months | 11.6 [2.0 to 30.7] | 40.0 [16.5 to 62.8] | 60.0 [12.6 to 88.2]
  24 months | 11.6 [2.0 to 30.7] | 40.0 [16.5 to 62.8] | 60.0 [12.6 to 88.2]

6. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of first dose of study treatment to the date of death due to any cause. Medians were estimated by the Kaplan-Meier method with 95% CIs estimated using the method of Brookmeyer and Crowley.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma: Participants with R/R non-GCB DLBCL received zanubrutinib plus rituximab for up to progressive disease or intolerance.
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Months | 11.20 [5.39 to 24.44] | NA [NA to NA] — NA = Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA = Not estimable due to insufficient number of participants with events

7. Secondary Outcome: OS: Survival Rate
Description: The OS was defined as the time from the date of first dose of study treatment to the date of death due to any cause. Survival rates were estimated by the Kaplan-Meier method with 95% CIs estimated using Greenwood's formula.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Relapsed/Refractory Follicular Lymphoma: Participants with R/R FL received zanubrutinib plus rituximab for up to progressive disease or intolerance.
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Percentage of Participants
  6 months | 72.7 [46.3 to 87.6] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  9 months | 55.9 [30.8 to 75.0] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  12 months | 44.7 [21.8 to 65.4] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  15 months | 33.6 [13.8 to 54.8] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  18 months | 33.6 [13.8 to 54.8] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events
  24 months | 33.6 [13.8 to 54.8] | 93.3 [61.3 to 99.0] | 100.0 [NA to NA] — NA = Not estimable due to insufficient number of participants with events

8. Secondary Outcome: Time To Response (TTR) As Determined By The Investigator
Description: The TTR was defined as the time from the date of the first dose of study treatment to the date of the first qualifying response (partial response or better).
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Relapsed/Refractory Marginal Zone Lymphoma: Participants with R/R MZL received zanubrutinib plus rituximab for up to progressive disease or intolerance.
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Months | 3.56 (2.054) | 6.15 (3.867) | 3.67 (1.631)

9. Secondary Outcome: Median TTR
Description: as for outcome 8
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Months | 2.79 [2.7 to 8.2] | 5.49 [2.6 to 13.8] | 2.73 [2.7 to 5.6]

10. Secondary Outcome: Complete Response Rate As Determined By The Investigator
Description: The percentage of participants whose best overall response met complete response or complete metabolic response criteria among all participants are reported. The 95% CI was calculated with Clopper-Pearson method.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Percentage of Participants | 10.0 [1.2 to 31.7] | 18.8 [4.0 to 45.6] | 0.0 [0.0 to 52.2]

11. Secondary Outcome: Number Of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) And Serious TEAEs
Description: A treatment-emergent adverse event was defined as an adverse event with an onset or worsening (if present pretreatment) starting on or after the first dose of study drug up to 30 days after discontinuation of zanubrutinib or 90 days after discontinuation of rituximab, whichever occurred later; or initiation of new anticancer therapy if it occurred prior to the other 2 dates. Worsening of a treatment-emergent adverse event to Grade 5 beyond Day 30 after the last dose of zanubrutinib or Day 90 after the last dose rituximab was also considered a treatment-emergent adverse event if the event occurred prior to initiation of new anticancer therapy.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
Number analyzed (Participants) | 20 | 16 | 5
Participants
  Participants With at Least 1 TEAE | 20 | 16 | 5
  Serious TEAEs | 7 | 4 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through approximately 2.5 years
Description: Participants were assessed for adverse events throughput the study and Follow-up Visit (30 days after last dose of zanubrutinib, 90 days after the last dose of rituximab, whichever occurred later). After this period, only new adverse events that were believed to be related to study treatment were reported.
Arm/Group | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma | Relapsed/Refractory Follicular Lymphoma | Relapsed/Refractory Marginal Zone Lymphoma
All-Cause Mortality (participants affected / at risk) | 13/20 | 1/16 | 0/5
Serious Adverse Events (participants affected / at risk) | 7/20 | 4/16 | 0/5
Other Adverse Events (participants affected / at risk) | 19/20 | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma (N=20) | Relapsed/Refractory Follicular Lymphoma (N=16) | Relapsed/Refractory Marginal Zone Lymphoma (N=5)
Lymph gland infection (Infections and infestations) | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed/Refractory Non-germinal Center B-cell-like Diffuse Large B-cell Lymphoma (N=20) | Relapsed/Refractory Follicular Lymphoma (N=16) | Relapsed/Refractory Marginal Zone Lymphoma (N=5)
White blood cell count decreased (Investigations) | 5 | 5 | 3
Neutrophil count decreased (Investigations) | 4 | 4 | 3
Alanine aminotransferase increased (Investigations) | 3 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1
Platelet count decreased (Investigations) | 3 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 1
Blood urine present (Investigations) | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4
Pneumonia (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 2
Asthenia (General disorders) | 0 | 1 | 2
Oedema peripheral (General disorders) | 1 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 2
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03520920/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT03520920/SAP_001.pdf